CLINICAL TRIAL: NCT02624102
Title: Efficacy of Trial-based Cognitive Therapy and Behavioral Activation in Treatment of Depression: a Randomized Clinical Trial
Brief Title: Efficacy of Trial-Based Cognitive Therapy and Behavioral Activation in Treatment of Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hemanny, Curt, M.D. (Individual)
Collaborators: Federal University of Bahia (Other)
Responsible Party: Principal Investigator, Curt Hemanny, Principal Investigator, Hemanny, Curt, M.D.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAAE 44663315.4.0000.5662
Record Dates: First submitted 2015-12-02; First posted 2015-12-08 (Estimated); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder; Cognitive behavioral therapy; Trial based cognitive therapy; Behavioral activation
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Antidepressive Agents; Drug Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cognitive therapy (Experimental): Major depressive disorder treated with cognitive therapy (Trial Based Cognitive Therapy plus Drug).
  Interventions: Behavioral: Trial based cognitive therapy
- Behavioral Therapy (Experimental): Major depressive disorder treated with behavioral therapy (Behavioral Activation plus drug).
  Interventions: Behavioral: Behavioral Activation
- Antidepressants (Other): Major depressive disorder treated only with antidepressants (Drug alone).
  Interventions: Drug: Antidepressants

INTERVENTIONS:
Behavioral: Trial based cognitive therapy — Patients with MDD, in use of antidepressants plus Trial Based Cognitive Therapy
  Other Names: TBCT
  Arms: Cognitive therapy
Behavioral: Behavioral Activation — Patients with MDD, in use of antidepressants plus Behavioral Activation
  Other Names: BA
  Arms: Behavioral Therapy
Drug: Antidepressants — Patients with MDD, in use of antidepressants (fluoxetine, citalopram, escitalopram, bupropion, etc.) without psychotherapy.
  Other Names: Pharmacotherapy, Control
  Arms: Antidepressants

SUMMARY:
Major Depressive Disorder (MDD) is a mood disorder, highly prevalent in Brazil and in world. The treatments of choice are the psychotropic drugs of the class of antidepressants and Behavioral or Cognitive Behavior Therapy (CBT). The aim of this study is to compare the efficacy of Trial Based Cognitive Therapy with the Behavioral Activation and pharmacotherapy in the treatment of MDD in a randomized clinical trial witch 96 patients with MDD,

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) is a mood disorder, highly prevalent in Brazil and in world. MDD is associated with an impaired quality of life and socio occupational functions. The treatments of choice are the psychotropic drugs of the class of antidepressants and Cognitive Behavior Therapy (CBT). Some of the patients with pharmacotherapy alone still symptomatic. This explains the association between psychotherapy and pharmacotherapy. The CBT seek to modify thoughts, emotions and behaviors and have shown efficacy in several mental disorders, including MDD. Among the CBT models, there is an emphasis on interventions that emphasize: 1) the modification or restructuring of thoughts and beliefs. In this point, the Trial based cognitive Therapy (TBCP) is an approach with a particular emphasis on the modification of core beliefs ; 2) the direct modification of behavior, such as the behavioral activation (BA) that analyzes contingencies and encourages the implementation of activities to improve mood. This project aims to compare the efficacy of TBCP with the BA in the treatment of MDD. For this, a randomized clinical trial will be conducted to treat 96 patients with MDD who are in drug treatment, which will be drawn to the interventions of TBCP most psychiatric drugs, BA more psychiatric drugs or pharmacotherapy alone, each group with 32 patients. Patients will be evaluated with scales and inventories to assess depression, quality of life and social functioning, and the data will be statistically compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Major Depressive Disorder
* Both Genres
* Minimum of 20 in BDI Score
* Refractory depressive disorder

Exclusion Criteria:

* Bipolar disorder
* High risk of suicide
* Borderline personality

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2015-09; Primary Completion 2017-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Severity of Depression | Twelve weeks (three months)
  Change from baseline in severity of depression at twelve weeks. Scale used is Beck Depression Inventory (BDI).

SECONDARY OUTCOMES:
WHOQoL | Twelve weeks (three months).
  Change from baseline in quality of life at twelve weeks. The scale used is World Health Organization Quality-of-Life Scale (WHOQoL-brief)
WHOQoL | One year.
  Change from baseline in quality of life at one year (follow-up). The scale used is World WHOQoL-brief.
Cognitive Distortions | Twelve weeks (Three months).
  Change from baseline in Cognitive Distortions at twelve weeks. The scale used is Cognitive Distortions Questionnaire (CD-Quest).
Cognitive Distortions | One year.
  Change from baseline in Cognitive Distortions at one years (follow-up). The scale used is CD-Quest.
Disability | twelve weeks.
  Change from baseline in Disability at twelve weeks). The scale used is Sheehan Disability Scale.
Disability | One year.
  Change from baseline in Disability at one year (follow-up). The scale used is Sheehan Disability Scale..
Severity of Depression (BDI) | One year.
  Change from baseline in Disability at one year (follow-up). Scale used is BDI.
Severity of Depression | One year.
  Change from baseline in severity of depression at one year (follow-up). Scale used is Hamilton Rating Scale for Depression (HRSD).
Severity of Depression (HRSD) | Twelve weeks.
  Change from baseline in severity of depression at twelve weeks. Scale used is HRSD.

CONTACTS AND LOCATIONS:
Overall Officials: Irismar Reis de Oliveira, Ph.D, Study Director — Federal University of Bahia
Locations (1):
- Curt Hemanny, Salvador, Estado de Bahia, Brazil